CLINICAL TRIAL: NCT01564914
Title: A Phase 2 Evaluation of TRC105 In Combination With Bevacizumab for the Treatment Of Recurrent or Progressive Glioblastoma That Has Progressed on Bevacizumab
Brief Title: A Phase 2 Evaluation of TRC105 In Combination With Bevacizumab in Patients With Glioblastoma
Acronym: 105GM201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Collaborators: The Cleveland Clinic (Other); Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105GM201/Case 1312
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — carotuximab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: A total of 6 initial patients were treated with 10 mg/kg of TRC105 monotherapy. All patients progressed within 2 months of initiating treatment, reflecting the rapid progression. Due to the lack of activity in this disease setting with TRC105 alone, the study was amended to treat patients with 10 mg/kg TRC105 weekly in combination with 10 mg/kg bevacizumab every two weeks.
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRC105, Bevacizumab (Experimental): Single arm study
  Interventions: Drug: TRC105; Drug: Bevacizumab

INTERVENTIONS:
Drug: TRC105 — 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
  Other Names: carotuximab
Drug: Bevacizumab — IV
  Other Names: Avastin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of TRC105 in patients with recurrent or progressive glioblastoma after prior antiangiogenic therapy (including anti-VEGF therapy)

DETAILED DESCRIPTION:
Angiogenesis plays a central role in the progression of solid cancer. TRC105 is an antibody to CD105, an important non-VEGF angiogenic target on proliferating endothelial cells. TRC105 inhibits angiogenesis, tumor growth and metastases in preclinical models. TRC105 has been well tolerated in patients with glioblastoma (GBM) as a single agent. The combination of TRC105 in combination with bevacizumab has demonstrated activity in bevacizumab refractory cancer patients. We hypothesize that TRC105 when administered with bevacizumab will have activity in GBM patients who progress on bevacizumab. By targeting a non-VEGF pathway, TRC105 has the potential to complement VEGF inhibition by bevacizumab, which could represent a major advance in GBM therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed glioblastoma, recurrent after prior external-beam fractionated radiotherapy and temozolomide chemotherapy.
2. Patients with documented radiographic progression following bevacizumab therapy for treatment of glioblastoma.
3. Patients with up to 3 prior recurrences are allowed.
4. Karnofsky performance status ≥ 70%.
5. Age ≥ 18 years old.
6. Normal organ function

Exclusion Criteria:

* Patients who have had previous treatment with TRC105.
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Patients with cirrhosis, or active viral or nonviral hepatitis.
* Patients with active bleeding or pathologic conditions that carry a high risk of bleeding,(i.e. hereditary hemorrhagic telangiectasia).
* Patients who are currently receiving anticoagulation treatment
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD PhD, Study Director — Tracon Pharmaceuticals Inc.
Locations (4):
- United States (4):
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened and enrolled at 4 sites
Groups:
- Carotuximab (TRC105), Bevacizumab: Single arm study
  Carotuximab (TRC105): 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
  Bevacizumab: IV 10 mg/kg every 2 weeks
- Carotuximab (TRC105): Single arm study
  Carotuximab (TRC105): 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
Period: Overall Study
Arm/Group | Carotuximab (TRC105), Bevacizumab | Carotuximab (TRC105)
Started | 16 | 6
Completed | 16 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who enrolled in the trial who received at least a portion of a dose were included
Groups:
- TRC105, Bevacizumab: Single arm study
  TRC105: 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
  Bevacizumab: IV 10 mg/kg every 2 weeks
- TRC105: Single arm
  TRC105: 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
- Total: Total of all reporting groups
Arm/Group | TRC105, Bevacizumab | TRC105 | Total
Number analyzed (Participants) | 16 | 6 | 22
Age, Customized [Median (Full Range); unit: years]
  Age | 64.5 [40 to 76] | 56.5 [38 to 73] | 62 [38 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 13 | 3 | 16
Screening Karnofsky Score [Number; unit: participants]
  Score = 60: requires occasional assistance | 1 | 3 | 4
  Score = 70: Can care for self; not normal activity | 4 | 0 | 4
  Score = 80: Normal activity with effort | 8 | 2 | 10
  Score = 90: Normal activities, minor symptoms. | 3 | 1 | 4
Cancer Histology [Count of Participants; unit: Participants]
  Glioblastoma | 15 | 5 | 20
  Giant Cell Glioblastoma | 1 | 0 | 1
  Astrocytoma | 0 | 1 | 1
Number of Prior Regimens [Median (Full Range); unit: prior regimens] | 2.5 [2 to 4] | 3 [1 to 5] | 3 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS)
Description: Overall survival assessed by determination from time of informed consent on trial to the date of death of each patient enrolled in the trial
Time Frame: 6 Months
Population: Patients treated with TRC105 and bevacizumab who expired. Overall survival was not captured in the monotherapy portion of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carotuximab (TRC105), Bevacizumab
Number analyzed (Participants) | 1
months | 5.75 [4.21 to 9.86]

2. Secondary Outcome: Median Duration That Patients Remained Progression Free on Study
Description: The median number of months that patients remained progression free was calculated using modified RANO criteria to determine progression. Modified RANO criteria is defined as follows: The largest cross-sectional area on the T1-weighted contrast-enhanced images was selected and measured in 2 dimensions with linear measures on the baseline MRI axial sequence. In addition, the largest cross-sectional area of a contiguous hyperintense lesion on FLAIR sequences was measured on the baseline MRI axial sequence. All subsequent scans were compared against these baseline measures (for both CE and FLAIR). New foci of FLAIR signal abnormality were recorded on each subsequent evaluation. Response was scored.
Time Frame: Patients are scanned every 8 weeks for approximately 6 months
Population: Patients with at least 1 on study scan were included in the efficacy population. The number of months that patients remained progression free was calculated for 5 evaluable monotherapy patients and 14 evaluable combination therapy patients.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carotuximab (TRC105), Bevacizumab: Single arm study
  Carotuximab (TRC105): 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
  Bevacizumab: IV
Arm/Group | Carotuximab (TRC105), Bevacizumab | Carotuximab (TRC105)
Number analyzed (Participants) | 14 | 5
months | 1.81 [1.25 to 2.07] | 1.38 [1.25 to 2.07]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse event frequency per patient according to CTCAE version 4.0.
Time Frame: Patients were followed for at least 28 days after the last dose of TRC105 study drug for adverse events, an average of 4 months
Population: Patients who received at least a portion of a dose of TRC105 and/or Bevacizumab
Measure: Count of Participants; unit: Participants
Groups:
- Carotuximab (TRC105), Bevacizumab: Single arm study
  Carotuximab (TRC105): 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
  Bevacizumab: IV 10 mg/kg every two weeks
Arm/Group | Carotuximab (TRC105), Bevacizumab | Carotuximab (TRC105)
Number analyzed (Participants) | 16 | 6
Participants
  Total SAEs | 6 | 3
  TRC105 Related SAEs | 2 | 0

4. Secondary Outcome: Number of Patients Who Respond to Study Treatment According to Modified RANO Criteria (Objective Response Rate (ORR)).
Description: Number of patients who respond to study treatment according to modified RANO criteria was calculated (Objective Response Rate (ORR)). Modified RANO criteria is defined as follows: The largest cross-sectional area on the T1-weighted contrast-enhanced images was selected and measured in 2 dimensions with linear measures on the baseline MRI axial sequence. In addition, the largest cross-sectional area of a contiguous hyperintense lesion on FLAIR sequences was measured on the baseline MRI axial sequence. All subsequent scans were compared against these baseline measures (for both CE and FLAIR). New foci of FLAIR signal abnormality were recorded on each subsequent evaluation. Response was scored.
Time Frame: Patients are scanned every 8 weeks
Population: Nineteen patients had measurable disease at baseline and received at least one follow up scan and were evaluable for the secondary efficacy outcome measure of PFS by modified RANO criteria. None of the patients treated on this study had a reduction in tumor burden compared to baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Carotuximab (TRC105) Alone: TRC105 alone 10 mg/kg weekly by intravenous administration on Days 1, 8, 15 and 22 of each 28-day cycle
Arm/Group | Carotuximab (TRC105), Bevacizumab | Carotuximab (TRC105) Alone
Number analyzed (Participants) | 16 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients were followed for at least 28 days after the last dose of TRC105 study drug for adverse events (on average 4 months).
Arm/Group | Carotuximab (TRC105), Bevacizumab | Carotuximab (TRC105)
All-Cause Mortality (participants affected / at risk) | 1/16 | 1/6
Serious Adverse Events (participants affected / at risk) | 6/16 | 3/6
Other Adverse Events (participants affected / at risk) | 16/16 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotuximab (TRC105), Bevacizumab (N=16) | Carotuximab (TRC105) (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 1 (1)
Peripheral Oedema (General disorders) | 1 (1) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 2 (2)
Mental Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotuximab (TRC105), Bevacizumab (N=16) | Carotuximab (TRC105) (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0)
Optic Neuropathy (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Breath Odour (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Defeacation Urgency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal Incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival Pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Oral Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Tooth Impacted (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 4 (4) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 12 (15) | 5 (5)
Feeling Hot (General disorders) | 1 (1) | 0 (0)
Gait Disturbance (General disorders) | 6 (8) | 0 (0)
Infusion Site Extravasation (General disorders) | 2 (2) | 0 (0)
Localised Oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Mucosal Inflammation (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 2 (5) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Back Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (6) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Cardiac Murmur (Investigations) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 1 (2) | 0 (0)
Lipase Increased (Investigations) | 1 (2) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Protein Total Decreased (Investigations) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 2 (4) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (13) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Amnesia (Nervous system disorders) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 2 (4) | 4 (5)
Apraxia (Nervous system disorders) | 1 (1) | 0 (0)
Balance Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Clumsiness (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 5 (6) | 2 (3)
Convulsion (Nervous system disorders) | 4 (4) | 3 (3)
Coordination Abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in Attention (Nervous system disorders) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 4 (5) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (15) | 3 (10)
Hemianopia Homonymous (Nervous system disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Loss of Proprioception (Nervous system disorders) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 2 (2) | 1 (1)
Mental Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Neurological Symptom (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 0 (0)
VIIth Nerve Paralysis (Nervous system disorders) | 2 (2) | 1 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Flat Affect (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Bilirubinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 0 (0)
Epistaxis (Vascular disorders) | 11 (14) | 1 (1)
Flushing (Vascular disorders) | 3 (3) | 0 (0)
Gingival Bleeding (Vascular disorders) | 4 (4) | 1 (1)
Haemoptysis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Telangiectasia (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less